CLINICAL TRIAL: NCT03553927
Title: Investigating the Physiological Effects of Weight Loss on Male Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18HH4412
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Male Infertility; Obesity; Weight Loss
Keywords: Male Infertility; Obesity
MeSH Terms: conditions — Infertility, Male; Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: 2 sub-studies Study A (men with a normal sperm concentration) Study B (men with a low sperm concentration)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Energy Diet (Other): Commercially available diet products
  Interventions: Dietary Supplement: Low Energy Diet
- NHS advice on healthy eating (Other): Dietary / lifestyle advice programme
  Interventions: Other: NHS advice on healthy eating

INTERVENTIONS:
Dietary Supplement: Low Energy Diet — Caloric restriction to achieve weight loss
  Arms: Low Energy Diet
Other: NHS advice on healthy eating — Advice on energy requirements as per the British Dietetic Association
  Arms: NHS advice on healthy eating

SUMMARY:
The purpose of this study is to determine the physiological effects of weight loss on seminal parameters in male participants with reduced reproductive capacity. Learning more about the physiological role of weight loss on reproductive function and metabolic profile of overweight and obese men may give us a better understanding of male fertility and improve the management of patients with reduced fertility. The effects of weight loss on seminal quality are not well understood.

DETAILED DESCRIPTION:
Participants will receive dietary supplements or National Health Service (NHS) advice on healthy eating to achieve weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 30 kg/m^2 [Part: 1, 2& 3]
* Evidence of reduced reproductive capacity (e.g. reduced sperm concentration [applicable for study B]

Exclusion Criteria:

* History of undescended testes, testicular surgery or mumps infection
* Hormonal therapy such as testosterone or selective oestrogen receptor modulators
* History of systemic cytotoxic therapy or pelvic radiotherapy
* Chronic systemic disease, such as cardiac, renal or liver failure
* At least one of the following:

Alcohol intake >30 units per week Smoking daily Recreational drug use at a frequency not less than weekly

* Acute illness likely to affect the result of study
* Impaired ability to provide full consent to take part in the study
* An occupation requiring strenuous physical exercise that may require a high energy diet

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 73 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channa Jayasena, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Healthcare Trust, North West London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sermondade N, Faure C, Fezeu L, Shayeb AG, Bonde JP, Jensen TK, Van Wely M, Cao J, Martini AC, Eskandar M, Chavarro JE, Koloszar S, Twigt JM, Ramlau-Hansen CH, Borges E Jr, Lotti F, Steegers-Theunissen RP, Zorn B, Polotsky AJ, La Vignera S, Eskenazi B, Tremellen K, Magnusdottir EV, Fejes I, Hercberg S, Levy R, Czernichow S. BMI in relation to sperm count: an updated systematic review and collaborative meta-analysis. Hum Reprod Update. 2013 May-Jun;19(3):221-31. doi: 10.1093/humupd/dms050. Epub 2012 Dec 12. PMID 23242914

RESULTS

PARTICIPANT FLOW:
Period: Study A (Men With a Normal Sperm Conc.)
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Study B (Men With a Low Sperm Conc.)
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Started | 22 | 23
Completed | 20 | 23
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Categorical [Count of Participants; unit: Participants] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  Participants
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration): <=18 years | 0 | 0 | 0
    Study A (men with a normal sperm concentration): Between 18 and 65 years | 12 | 12 | 24
    Study A (men with a normal sperm concentration): >=65 years | 0 | 0 | 0
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration): <=18 years | 0 | 0 | 0
    Study B (men with a low sperm concentration): Between 18 and 65 years | 20 | 23 | 43
    Study B (men with a low sperm concentration): >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  Years
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 40.2 (9.6) | 39.4 (6.4) | 39.8 (8)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 37.7 (6.6) | 39.5 (7.5) | 38.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 35 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 22 | 39
  Mixed | 0 | 2 | 2
  Asian | 7 | 9 | 16
  Black | 0 | 1 | 1
  Arab | 6 | 1 | 7
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 35 | 67
Weight [Mean (Standard Deviation); unit: Kilograms] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  Kilograms
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 109.5 (10.8) | 114.1 (11) | 112.6 (11.4)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 116.8 (17.3) | 117 (21.9) | 116.9 (19.7)
Waist circumference [Mean (Standard Deviation); unit: Centimetres] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  Centimetres
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 117.3 (7.6) | 119.5 (9.1) | 118.8 (8.4)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 123.4 (9.7) | 120.9 (12.9) | 122.1 (11.5)
Sperm concentration [Mean (Standard Deviation); unit: million sperms/mL] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  million sperms/mL
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 38.3 (15) | 54.2 (21.3) | 46.2 (19.8)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 5.3 (3.4) | 9.8 (10.0) | 7.6 (7.9)
Semen volume [Mean (Standard Deviation); unit: ml] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  ml
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 3.3 (1.4) | 3.9 (1.1) | 3.6 (1.3)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 3.7 (1.8) | 3.3 (1.4) | 3.4 (1.6)
Progressive motility [Mean (Standard Deviation); unit: percentage of progressively motile sperm] — This type of motility refers to sperm that swim progressively, mostly in a straight line or large circles Population: The overall number of baseline participants refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure progressive motility.
  percentage of progressively motile sperm
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 41 (16) | 45 (8) | 43 (12)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 20 | 39
    Study B (men with a low sperm concentration) | 28.7 (13.2) | 33.4 (14.5) | 31.1 (13.9)
Total motility [Mean (Standard Deviation); unit: percentage of sperm that is motile] — Total motility refers to the percentage of sperm making any sort of movement. Population: The overall number of baseline participants refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure total motility.
  percentage of sperm that is motile
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 48 (17) | 52 (8) | 50 (13)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 20 | 39
    Study B (men with a low sperm concentration) | 35 (13.8) | 40 (15.5) | 36 (15)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  kg/m^2
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 35.3 (4.1) | 36.2 (2.4) | 35.8 (3.3)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 38 (4) | 38 (6.3) | 38 (5.3)
DNA Fragmentation Index [Mean (Standard Deviation); unit: percentage of sperm with fragmented DNA] — Percentage of sperm with fragmented DNA Population: The overall number of baseline participants refers to the total number after combining the two sub-studies Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure DNA Fragmentation Index..
  percentage of sperm with fragmented DNA
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 11.9 (13.1) | 15.9 (6.7) | 13.8 (9.5)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 12 | 17 | 29
    Study B (men with a low sperm concentration) | 15.8 (7.7) | 12.1 (9.5) | 13.6 (8.9)
Testosterone [Mean (Standard Deviation); unit: nmol/l] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  nmol/l
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 12.7 (4.2) | 12.3 (2.5) | 12.5 (3.4)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 12.6 (5.1) | 14.6 (5) | 13.4 (5.1)
Sex hormone-binding globulin (SHBG) [Mean (Standard Deviation); unit: nmol/l] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  nmol/l
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 21.8 (8.1) | 25.2 (8.7) | 23.5 (8.4)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 21.4 (10.6) | 24.8 (9.6) | 23.2 (10.1)
Reactive oxygen species (ROS) [Median (Inter-Quartile Range); unit: RLU/sec/million sperm] — ROS is measured by oxidative colour change of luminol per second per million sperm Population: ROS was only measured in Study B. Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure ROS.
  .
  RLU/sec/million sperm
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 0 | 0 | 0
    Study B (men with a low sperm concentration): number analyzed (Participants) | 13 | 17 | 30
    Study B (men with a low sperm concentration) | 8.6 [5.5 to 177] | 3.6 [1.2 to 37] | 7.1 [2 to 46]
Morphology [Mean (Standard Deviation); unit: percentage of sperm of normal morphology] — the percentage (%) of sperm that appear normal when semen is viewed under a microscope. Population: Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to analyze morphology.
  percentage of sperm of normal morphology
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 1.6 (1.3) | 1.8 (1.4) | 1.7 (1.3)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 17 | 20 | 37
    Study B (men with a low sperm concentration) | 0.4 (0.7) | 1 (0.8) | 0.7 (0.8)
Luteinizing Hormone (LH) [Mean (Standard Deviation); unit: IU/l] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  IU/l
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 3.2 (1) | 3.5 (1.7) | 3.3 (1.4)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 3.7 (0.9) | 4.3 (1.5) | 4 (1.2)
Follicle Stimulating Hormone (FSH) [Mean (Standard Deviation); unit: IU/l] — Population: The overall number of baseline participants refers to the total number after combining the two sub-studies
  IU/l
    Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12 | 24
    Study A (men with a normal sperm concentration) | 4.2 (2.6) | 4.4 (1.9) | 4.3 (2.8)
    Study B (men with a low sperm concentration): number analyzed (Participants) | 20 | 23 | 43
    Study B (men with a low sperm concentration) | 5.6 (2.9) | 5 (2.5) | 5.3 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Sperm Concentration
Description: The number of sperm per millimeter of semen. Sperm concentration is an important factor affecting male fertility. It is calculated on a standard semen analysis
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies
Measure: Mean (Standard Deviation); unit: million sperms/mL
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 32 | 35
million sperms/mL
  Study A (men with normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with normal sperm concentration) | 53.6 (36.4) | 58.5 (32.8)
  Study B (men with low sperm concentration): number analyzed (Participants) | 20 | 23
  Study B (men with low sperm concentration) | 20.1 (59.16) | 15 (16.8)

2. Secondary Outcome: Total Motility
Description: Total motility refers to the percentage of sperm making any sort of movement.
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure total motility.
Measure: Mean (Standard Deviation); unit: percentage of sperm that is motile
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 29 | 33
percentage of sperm that is motile
  men with a normal sperm concentration: number analyzed (Participants) | 12 | 12
  men with a normal sperm concentration | 59.5 (9.6) | 60.8 (6.3)
  men with a low sperm concentration: number analyzed (Participants) | 17 | 21
  men with a low sperm concentration | 48.9 (12) | 45.4 (16.1)

3. Secondary Outcome: Progressive Motility
Description: This type of motility refers to sperm that swim progressively, mostly in a straight line or large circles.
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure progressive motility.
Measure: Mean (Standard Deviation); unit: percentage of progressively motile sperm
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 29 | 33
percentage of progressively motile sperm
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 53.3 (10.4) | 53.9 (6.1)
  study B (men with a low sperm concentration): number analyzed (Participants) | 17 | 21
  study B (men with a low sperm concentration) | 42.8 (14.1) | 39.6 (17)

4. Secondary Outcome: DNA Fragmentation Index (DFI)
Description: Percentage of sperm with fragmented DNA
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure DNA fragmentation index.
Measure: Mean (Standard Deviation); unit: Percentage of sperm with fragmented DNA
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 24 | 29
Percentage of sperm with fragmented DNA
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 7.7 (8.7) | 19.8 (9.6)
  study B (men with a low sperm concentration): number analyzed (Participants) | 12 | 17
  study B (men with a low sperm concentration) | 18.4 (11.7) | 11.2 (11)

5. Secondary Outcome: Testosterone
Description: Testosterone is the primary androgen in men and is synthesized in the testes. It can be measured in the serum.
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies.
  One participant in Low Energy Diet arm in study B did not have this measurement due to insufficient sample.
Measure: Mean (Standard Deviation); unit: nmol/l
Groups:
- Low Energy Diet, Men With Normal Sperm Concentration: Commercially available diet products
  Low Energy Diet: Caloric restriction to achieve weight loss
- NHS Advice on Healthy Eating, Men With Normal Sperm Concentration: Dietary / lifestyle advice programme
  NHS advice on healthy eating: Advice on energy requirements as per the British Dietetic Association
Arm/Group | Low Energy Diet, Men With Normal Sperm Concentration | NHS Advice on Healthy Eating, Men With Normal Sperm Concentration
Number analyzed (Participants) | 31 | 35
nmol/l
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 13.6 (5) | 12.4 (2.8)
  study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 23
  study B (men with a low sperm concentration) | 15.6 (6.2) | 13.7 (4.1)

6. Secondary Outcome: Sex Hormone-Binding Globulin (SHBG)
Description: SHBG is a protein that is produced by the liver and binds tightly to the hormones testosterone, dihydrotestosterone (DHT) and oestradiol, and transports them in the blood in an inactive form.
Time Frame: 16 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 31 | 35
nmol/l
  (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  (men with a normal sperm concentration) | 30.2 (12.6) | 26.4 (7)
  study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 23
  study B (men with a low sperm concentration) | 24.2 (12.4) | 22.6 (8.1)

7. Secondary Outcome: Reactive Oxygen Species (ROS)
Description: ROS is measured by oxidative colour change of luminol per second per million sperm.
Time Frame: 16 weeks
Population: ROS was only measured in Study B. Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure ROS.
Measure: Median (Inter-Quartile Range); unit: RLU/sec/million sperm
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 14 | 19
RLU/sec/million sperm | 13 [3 to 39.1] | 5 [0.9 to 37.4]

8. Secondary Outcome: Morphology
Description: the percentage of sperm that appear normal when semen is viewed under a microscope
Time Frame: 16 weeks
Population: The overall number of participants analyzed refers to the total number after combining the two sub-studies.
  Some participants in Study B were not assessed for this measure due to sperm concentrations that were too low to measure morphology.
Measure: Mean (Standard Deviation); unit: percentage of sperm of normal morphology
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 27 | 31
percentage of sperm of normal morphology
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 1.2 (1.1) | 1.9 (1.7)
  Study B (men with a low sperm concentration): number analyzed (Participants) | 15 | 19
  Study B (men with a low sperm concentration) | 0.6 (0.6) | 1.3 (1.7)

9. Secondary Outcome: Luteinizing Hormone (LH)
Description: LH produced in the pituitary gland, stimulates the leydig cells in the testes to produce testosterone.
Time Frame: 16 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/l
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 31 | 35
IU/l
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 3.3 (1.4) | 2.8 (1.2)
  Study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 23
  Study B (men with a low sperm concentration) | 3.5 (1.4) | 3.7 (1.5)

10. Secondary Outcome: Follicle Stimulating Hormone (FSH)
Description: FSH produced in the pituitary gland, stimulates the testes to produce mature sperm.
Time Frame: 16 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/l
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
Number analyzed (Participants) | 31 | 35
IU/l
  Study A (men with a normal sperm concentration): number analyzed (Participants) | 12 | 12
  Study A (men with a normal sperm concentration) | 3.8 (2.1) | 4.5 (2.2)
  Study B (men with a low sperm concentration): number analyzed (Participants) | 19 | 23
  Study B (men with a low sperm concentration) | 5.4 (2.6) | 5 (2.4)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were monitored for as defined as per clinicaltrials.gov definitions.
Arm/Group | Low Energy Diet | NHS Advice on Healthy Eating
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03553927/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03553927/ICF_002.pdf